CLINICAL TRIAL: NCT00352118
Title: Phase II Pilot Study of TPF (Docetaxel, Cisplatin, and 5-FU) Induction Chemotherapy Followed by Concurrent Cisplatin and Reduced Dose Radiation in Locally Advanced Head and Neck Cancer
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Locally Advanced Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low dose radiation treatment was not appropriate for these patients.
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005LS012; UMN-0502M67486
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Head and Neck Cancer
Keywords: oral complications of radiation therapy; oral complications of chemotherapy; mucositis; xerostomia; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis; Xerostomia; Squamous Cell Carcinoma of Head and Neck | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Cisplatin; Docetaxel; Fluorouracil; Surgical Procedures, Operative; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy + Low Dose Radiation (Experimental): Patients receiving chemotherapy and Low Dose (60 Gy) Radiation per protocol.
  Interventions: Biological: filgrastim; Biological: pegfilgrastim; Drug: cisplatin; Drug: docetaxel; Drug: fluorouracil; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — subcutaneously on Days 5-14, repeating every 3 weeks for 2 courses.
  Other Names: G-CSF; Neupogen
Biological: pegfilgrastim — If applicable on day 5, repeating every 3 weeks for 2 courses.
  Other Names: Neulasta, G-CSF
Drug: cisplatin — Intravenous over 1 hour on day 1, every 3 weeks for 3 courses.
  Other Names: CDDP; cisplatinum; cis-diamminedichloridoplatinum; Platinol AQ
Drug: docetaxel — Intravenous over 1 hour on day 1.
  Other Names: Taxotere(R)
Drug: fluorouracil — Intravenous continuously on days 1-4.
  Other Names: 5-FU; 5-fluorouracil; Adrucil
Procedure: conventional surgery — As appropriate, neck dissection.
  Other Names: surgery
Radiation: radiation therapy — 60 Gy 5 days/week x 6 weeks with cisplatin
  Other Names: radiation

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, cisplatin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving combination chemotherapy together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with radiation therapy works in treating patients with locally advanced head and neck cancer. The doctor also wants to find out if patients who receive this treatment need a feeding tube 1 year after starting treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine feeding tube dependency at 12 months in patients with locally advanced head and neck cancer treated with induction chemotherapy comprising docetaxel, cisplatin, and fluorouracil followed by cisplatin and reduced-dose radiotherapy.

Secondary

* Determine the progression-free, disease-free, and overall survival of patients treated with this regimen.
* Determine the pattern of failure in patients treated with this regimen.
* Evaluate the quality of life of patients treated with this regimen.
* Assess pre- and post-treatment swallowing ability of patients and the impact on their quality of life.

Tertiary

* Quantify salivary flow rates of patients receiving chemotherapy with radiotherapy for head and neck malignancy.
* Evaluate the quality of saliva by examining total protein concentrations.
* Quantify proangiogenic cytokines (interleukin [IL]-1, IL-6, IL-8, and vascular endothelial growth factor) in the saliva of these patients.
* Determine the degree of mucositis and xerostomia of patients receiving chemotherapy with radiotherapy for head and neck malignancy.
* Compare salivary flow rates with the grade of mucositis and xerostomia of patients receiving chemotherapy with radiotherapy for head and neck malignancy.

OUTLINE: This is a pilot study.

* Induction therapy: Patients receive docetaxel IV over 1 hour and cisplatin IV over 1 hour on day 1 followed by fluorouracil IV continuously on days 1- 4. Patients also receive filgrastim (G-CSF) subcutaneously (SC) on days 5-14 or pegfilgrastim SC on day 5. Treatment repeats every 3 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving a partial or clinical complete response proceed to chemoradiotherapy 3 weeks later.
* Chemoradiotherapy: Patients receive cisplatin IV over 1 hour on day 1. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients also undergo concurrent reduced-dose radiotherapy 5 days a week for 6 weeks.
* Surgery: Approximately 6 to 8 weeks after completing chemoradiotherapy, patients with residual neck disease or disease initially staged at N2 or greater undergo neck dissection.

Saliva is collected periodically to measure flow rates and quality; quantify proangiogenic cytokines (interleukin [IL]-1, IL-6, IL-8 and vascular endothelial growth factor); and examine the grade of mucositis and xerostomia.

Quality of life is assessed at baseline, before chemoradiotherapy, 1 month after the last radiation treatment, every 3 months for 1 year, and then every 6 months for 1 year.

After completion of study treatment, patients are followed periodically for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * Stage IVA or IVB disease

    * Stage III disease allowed provided patient may benefit from organ preservation or patient refused surgery
* Measurable or evaluable disease
* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine ≤ 1.5 mg/dL OR glomerular filtration rate ≥ 60 mL/min
* Bilirubin normal
* Alkaline phosphatase (AP) and AST or ALT must be within the following ranges:

  * AP normal AND AST or ALT ≤ 5 times upper limit of normal (ULN)
  * AP ≤ 2.5 times ULN AND AST or ALT ≤ 1.5 times ULN
  * AP ≤ 5 times ULN AND AST or ALT normal

Exclusion Criteria:

* Salivary gland, sinus, or nasopharyngeal primary disease
* Evidence of distant metastatic disease
* Pregnant or nursing
* Positive pregnancy test (Fertile patients must use effective contraception during study treatment and for 3 months after completion of study treatment)
* Other malignancy within the past 5 years except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other malignancy in which stage and nature of disease is such that it is unlikely to affect survival for the next 3 years
* Peripheral neuropathy ≥ grade 2
* Hearing loss ≥ grade 2
* Severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 and/or cisplatin or other platinum analogs
* Poor nutritional status, in the opinion of the investigator
* Active infection
* Active ischemic heart disease
* Myocardial infarction within the past 6 months
* Prior radiotherapy above the clavicles
* Prior chemotherapy
* Prior surgery to the primary tumor except biopsy
* Concurrent amifostine or other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank G. Ondrey, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Masonic Cancer Center physicians' clinics.
Groups:
- Chemotherapy + Low Dose Radiation: Patients receiving combination chemotherapy plus low dose radiation
Period: Overall Study
Arm/Group | Chemotherapy + Low Dose Radiation
Started | 4
Completed | 0
Not Completed | 4
Not completed — Physician Decision | 4

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy + Low Dose Radiation
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Feeding Tube Dependency
Description: All patients were non-evaluable and study was terminated early. There is no measure of outcome.
Time Frame: at 12 months
Population: All patients were non-evaluable - did not receive radiation dose per protocol.
Arm/Group | Chemotherapy + Low Dose Radiation
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Days With Progression-free Survival
Description: All patients were non-evaluable and study was terminated early. There is no measure of outcome. Utilizing RECIST criteria.
Time Frame: Between date of registration to date of first treatment failure or death.
Population: All patients were non-evaluable - did not receive radiation dose per protocol.
Arm/Group | Chemotherapy + Low Dose Radiation
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Days - Overall Survival
Description: as for outcome 2
Time Frame: Between date of registration to date of death.
Population: All patients were non-evaluable - did not receive radiation dose per protocol.
Arm/Group | Chemotherapy + Low Dose Radiation
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Days With Disease Free Survival
Description: All patients were non-evaluable and study was terminated early. There is no measure of outcome. RECIST criteria measurement.
Time Frame: From Date of Registration to Date of First Treatment Failure or Death
Population: All patients were non-evaluable - did not receive radiation dose per protocol.
Arm/Group | Chemotherapy + Low Dose Radiation
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Treatment Failure
Description: All patients were non-evaluable and study was terminated early. There is no measure of outcome. Measure using RECIST criteria.
Time Frame: Number of Days from Complete or Partial Response to First Date of Recurrence or Progression
Population: All patients were non-evaluable - did not receive radiation dose per protocol.
Arm/Group | Chemotherapy + Low Dose Radiation
Number analyzed (Participants) | 0

6. Secondary Outcome: Swallowing Ability - Quality of Life Scores
Description: All patients were non-evaluable and study was terminated early. There is no measure of outcome. Utilizing Swallowing Portion of ASHA Functional Communication Measure for Swallowing (FCM) and Dysphagia Outcome and Severity Scale (DOSS).
Time Frame: Baseline, before chemoradiation, 30 days after last radiation treatment, every 3 months for the first year, then every 6 months for year 2.
Population: All patients were non-evaluable - did not receive radiation dose per protocol.
Arm/Group | Chemotherapy + Low Dose Radiation
Number analyzed (Participants) | 0

7. Secondary Outcome: Quality of Life (QOL) by Functional Assessment of Cancer Therapy-H&N QOL Questionnaire
Description: All patients were non-evaluable and study was terminated early. There is no measure of outcome.
Time Frame: baseline, before chemoradiotherapy, 1 month after the last radiation treatment, every 3 months for 1 year, and then every 6 months for 1 year
Population: All patients were non-evaluable - did not receive radiation dose per protocol.
Arm/Group | Chemotherapy + Low Dose Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Chemotherapy + Low Dose Radiation
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
All 4 patients received high dose radiation (66-70 Gy). The radiation oncologist on this study deemed low dose radiation treatment was not appropriate for these patients. Therefore, the study participants are not evaluable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes